CLINICAL TRIAL: NCT06737692
Title: Investigation of the Effects of Aerobic and Resistance Exercise Training in Individuals with Gastrointestinal Cancer and Cachexia: Randomized Controlled Single-Blind Study
Brief Title: Effects of Aerobic and Resistance Exercise Training in Individuals with Cancer Cachexia
Acronym: Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Didem KARADIBAK, Director, Head of Cardiopulmonary Physiotherapy, Principal Investigator, Clinical Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEUFTR-ERGIN-001
Record Dates: First submitted 2024-12-02; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-10

CONDITIONS: Cancer Cachexia (CC)
Keywords: exercise; cancer; cachexia; aerobic; resistance
MeSH Terms: conditions — Motor Activity; Neoplasms; Cachexia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A total of 40 participants aged 18 to 65, diagnosed with gastrointestinal cancer and cachexia, will be included in the study. Participants will be randomly assigned to the exercise group (aerobic and resistance training) or the control group (standard care), with 20 individuals in each group. The study will be single-blind, meaning the Outcomes Assessor will not know which group the participants belong to.
Who Masked: Outcomes Assessor
Masking Description: The study will be single-blind, meaning that the Outcomes Assessor and the researcher implementing the exercise program will be different individuals. The Outcomes Assessor will not be aware of which group the participants belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): The exercise group will participate in a supervised and home-based exercise program consisting of aerobic and resistance exercises over 12 weeks.
  Supervised Aerobic Exercises: Conducted every two weeks, 3 days/week (on days 11-13 post-systemic treatment). The supervised aerobic exercises will consist of 20 minutes on a treadmill at a heart rate corresponding to 55-75% of the Karvonen formula. Warm-up and cool-down will be performed at 30-40% of the Karvonen heart rate for 5 minutes.
  Supervised Resistance Exercises: Conducted every 2 weeks on consecutive days (days 11 and 13 post-systemic treatment). Resistance training will involve 12 different exercises targeting major muscle groups, using body weight and resistance bands, at an effort level of 5-7 on the Borg scale, with 8-12 repetitions and 1-3 sets.
  On weeks without supervised exercises, participants will follow a home exercise program that includes breathing exercises, walking for 20-30 minutes, and resistance exercises.
  Interventions: Other: Exercise
- Control group (No Intervention): Participants in the control group will be instructed to maintain their daily lifestyle, including physical activity, during their participation in the study. After completion of the study, participants in the control group will be offered a supervised aerobic and resistance exercise program and will be administered the same exercise program.

INTERVENTIONS:
Other: Exercise — Supervised Aerobic Exercises: Conducted every two weeks, three days a week (on days 11-13 post-systemic treatment). The supervised aerobic exercises will consist of 20 minutes on a treadmill at a heart rate corresponding to 55-75% of the Karvonen formula. Warm-up and cool-down will be performed at 30-40% of the Karvonen heart rate for 5 minutes.
  Supervised Resistance Exercises: Conducted every two weeks on consecutive days (days 11 and 13 post-systemic treatment).
  Resistance training will involve 12 different exercises targeting major muscle groups, using body weight and resistance bands, at an effort level of 5-7 on the Borg scale, with 8-12 repetitions and 1-3 sets. The intensity will be progressively adjusted based on the individual's perceived exertion.
  On weeks without supervised exercises, participants will follow a home exercise program that includes breathing exercises, walking for 20-30 minutes, and resistance exercises.
  Arms: Exercise group

SUMMARY:
This study aims to evaluate the effects of a 12-week aerobic and resistance exercise program in cancer patients with cachexia compared to standard care.

A total of 40 participants aged 18 to 65, diagnosed with gastrointestinal cancer and cachexia, will be included in the study. Participants will be randomly assigned to the exercise group (aerobic and resistance training) or the control group (standard care), with 20 individuals in each group.

Before the 12-week intervention, both the exercise and control groups will undergo evaluations. Demographic and clinical data will be recorded. The following assessments will be conducted:

Body Composition: Bioelectrical impedance analysis Sarcopenia Assessment: SARC-F questionnaire Functional Exercise Capacity: 6-minute walk test Gait Parameters: 8-meter walk test Mobility and Balance: Timed Up and Go test Muscle Strength: Knee extensor and hand grip strength measured with dynamometers 30-second sit-to-stand test Additionally, participants will complete several questionnaires, including the Edmonton Symptom Assessment Scale, Karnofsky Performance Status scale, FRAIL scale, Fatigue Severity Scale, and EORTC-QLQ30.

The exercise group will participate in a supervised and home-based exercise program consisting of aerobic and resistance exercises over 12 weeks.

The intensity will be progressively adjusted based on the individual's perceived exertion.

DETAILED DESCRIPTION:
Cancer cachexia is a multifactorial syndrome characterized by progressive functional impairment and loss of skeletal muscle mass, which does not improve with nutritional support. This study aims to evaluate the effects of a 12-week aerobic and resistance exercise program in cancer patients with cachexia compared to standard care.

A total of 40 participants aged 18 to 65, diagnosed with gastrointestinal cancer and cachexia, will be included in the study. Participants will be randomly assigned to the exercise group (aerobic and resistance training) or the control group (standard care), with 20 individuals in each group.

The study will be single-blind, meaning the outcome assessor will not know which group the participants belong to.

Before the 12-week intervention, both the exercise and control groups will undergo evaluations. Demographic and clinical data will be recorded. The following assessments will be conducted:

Body Composition: Bioelectrical impedance analysis Sarcopenia Assessment: SARC-F questionnaire Functional Exercise Capacity: 6-minute walk test Gait Parameters: 8-meter walk test Mobility and Balance: Timed Up and Go test Muscle Strength: Knee extensor and hand grip strength measured with dynamometers 30-second sit-to-stand test Additionally, participants will complete several questionnaires, including the Edmonton Symptom Assessment Scale, Karnofsky Performance Status scale, FRAIL scale, Fatigue Severity Scale, and EORTC-QLQ30.

The exercise group will participate in a supervised and home-based exercise program consisting of aerobic and resistance exercises over 12 weeks.

Supervised Aerobic Exercises: Conducted every two weeks, three days a week. Supervised Resistance Exercises: Conducted every two weeks on consecutive days. On weeks without supervised exercises, participants will follow a home exercise program that includes breathing exercises, walking for 20-30 minutes, and resistance exercises.

The supervised aerobic exercises will consist of 20 minutes on a treadmill at a heart rate corresponding to 55-75% of the Karvonen formula. Warm-up and cool-down will be performed at 30-40% of the Karvonen heart rate for 5 minutes.

Resistance training will involve 12 different exercises targeting major muscle groups, using body weight and resistance bands, at an effort level of 5-7 on the Borg scale, with 8-12 repetitions and 1-3 sets.

The intensity will be progressively adjusted based on the individual's perceived exertion.

ELIGIBILITY:
Inclusion Criteria:

* Stage III-IV gastrointestinal cancer diagnosis
* Age 18-65
* Receiving systemic treatment (chemotherapy and/or targeted therapy and/or immunotherapy), at least 6 weeks after surgery,
* Karnofsky performance score 80 and above,
* Diagnosis of cachexia according to diagnostic criteria and Glasgow Prognostic Score (5,30) (>5% weight loss in the last 6 months or >2% weight loss in patients with BMI less than 20 kg/m2 or >2% weight loss in sarcopenic individuals)

Exclusion Criteria:

* Musculoskeletal disorder
* Neurological disorder
* Severely impaired hematological capacity
* History of cardiac disease
* Uncontrolled hypertension
* Severe renal insufficiency
* Advanced osteoporosis
* Decreased ability to stand or walk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Demographic and Clinical Information | At baseline and after 12 weeks of exercise training
  Age, gender, occupation, education status, marital status, medical history, family medical history, medications used, smoking and exercise habits, clinical information about cancer (diagnosis date, cancer stage, treatment received, and treatment start and end times) will be recorded.
Weight Assessment | At baseline and after 12 weeks of exercise training
  Weight change in a certain period and percentage of initial weight are used to determine weight loss. Weight loss of 5%, 10% or 20% in a certain period is associated with an increased risk of malnutrition. The participants' weights will be recorded in kilograms.
Height Assessment | At baseline and after 12 weeks of exercise training
  The participants' heights will be recorded in centimeters.
Body Mass Index Assessment Body Mass Index Assessment | At baseline and after 12 weeks of exercise training
  The participants' Body Mass Index (BMI) values will be recorded in kg/m² (kilograms per square meter).
Assessment of Muscle Strength | At baseline and after 12 weeks of exercise training
  Quadriceps femoris muscle strength will be evaluated using a digital dynamometer (Lafayette, USA). The tests will be performed in the sitting position. Muscle strength will be tested in the middle of the joint range of motion, and the maximum isometric contraction will be measured for 5 seconds. The muscle strength measurement will be repeated 3 times on the right and left sides, and the best value obtained will be recorded in kilograms (kg).
  Hand grip strength will be measured with a hydraulic dynamometer (Jamar, Sammons Preston Rolyan, Chicago, USA). The test will be performed while patients are sitting comfortably with the shoulder adducted, the forearm neutrally rotated, the elbow flexed 90° and the forearm and wrist in a neutral position. Patients will be instructed to perform a maximum isometric contraction. The participants' hand grip strengths will be recorded in kilograms.
Assessment of Lower Extremity Performance | At baseline and after 12 weeks of exercise training
  Lower extremity performance will be evaluated with a 30-second sit-to-stand test, in which the number of times a person can sit down and stand up in 30 seconds is recorded.
Sarcopenia Assessments | At baseline and after 12 weeks of exercise training
  The steps determined by ESWGOP will be followed in sarcopenia screening. The 5-question SARC-F questionnaire is a rapid screening questionnaire used in sarcopenia assessment. Responses are scored between 0-2 and the total score is between 0-10. A total score of 4 or more indicates the presence of a risk for sarcopenia.
Assessment of Muscle and Fat Mass | At baseline and after 12 weeks of exercise training
  Bioelectrical impedance analysis (Inbody 720) will be used for muscle and fat mass assessment. Participants' muscle and fat mass will be recorded in kilograms.
Mobility, balance and performance assessment | At baseline and after 12 weeks of exercise training
  For mobility, balance and performance assessment; Timed Up and Go test (TUG) will be used. TUG will be performed by standing up from a chair (sitting height 46 cm), walking 3 m to a line marked on the floor, crossing the line, turning around and walking back, and sitting on a chair.
  For TUG-cognitive, the individual will be instructed to count backwards by 3 from a random number between 20 and 100 while completing the TUG. The number will be given immediately after the researcher says "go", and errors in subtraction will not be corrected.
  In TUG-manual, the individual will be asked to pick up and carry a glass full of beans without spilling while completing the TUG. The glass will be placed on a solid surface 90° to the right of the individual while they are sitting, and they will be asked to put the glass back in the same spot before sitting down again.
Assessment of Functional Exercise Capacity | At baseline and after 12 weeks of exercise training
  A 6-minute walk test (6 MWT) will be used to assess functional exercise capacity. Participants will be asked to walk as fast as possible on a 30-meter straight corridor in the 6 MWT and the distance covered will be recorded in meters. During 6 MWT, walking distance, speed and cadence will be assessed using a wireless motion detection device (G-Walk, BTS Bioengineering SpA, Italy) attached to the individual's waist using a semi-elastic belt over L4-L5.
Assessment of Gait Parameters | At baseline and after 12 weeks of exercise training
  Individuals will be asked to walk as naturally as possible along an 8-meter path at a speed of their own choosing to assess the time-distance parameters of walking. The 8-meter walk test will measure the time-distance parameters of gait, including step length, stance and swing phases, single support and double support phases. During 8-meter walk test, walking distance, speed, cadence and time-distance parameters of gait will be assessed using a wireless motion detection device (G-Walk, BTS Bioengineering SpA, Italy) attached to the individual's waist using a semi-elastic belt over L4-L5.

SECONDARY OUTCOMES:
Performance Assessment | At baseline and after 12 weeks of exercise training
  Functional status will be assessed using the Karnofsky Performance Status (KPD) scale. It is considered the gold standard of performance measurement for cancer patients. Individuals will rate their functional status using the KPD scale, which ranges from 30 (I feel severely disabled and need to be hospitalized) to 100 (I feel normal; I have no complaints or symptoms). In the literature, it is generally accepted that individuals who score 70 points and above have adequate functional status. This score indicates that the individual is at a level where they can care for themselves, but their normal activity has decreased and they are unable to do active work.
Evaluation of Symptoms | At baseline and after 12 weeks of exercise training
  The Edmonton Symptom Assessment Scale will be used to evaluate the symptoms of participants in both groups. The symptoms included in the scale are pain, fatigue, drowsiness, nausea, loss of appetite, dyspnea, depression, anxiety, feeling unwell and other problems. The severity of each symptom is scored between 0 and 10. A score of 0 indicates no symptoms, while a score of 10 indicates that the symptom is felt very severely.
Frailty Assessment | At baseline and after 12 weeks of exercise training
  Morley et al. found that the five-item 'FRAIL Scale' was effective in detecting frailty. In addition to the patient's general health status, the questionnaire evaluates with questions about comorbidities; patients receive zero or one point according to the answer given for each question. A total of 0 is considered normal (non-frail), 1-2 is pre-frail and a score of >2 is frail. The validity and reliability of the questionnaire in Turkish was demonstrated by Hymabaccus et al. in 2017.
Assessment of Cancer-Related Fatigue | At baseline and after 12 weeks of exercise training
  The Fatigue Severity Scale (FSS) will be used to assess the participants' level of cancer-related fatigue. FSS is a scale consisting of 9 questions that assess fatigue. Each item is scored between 0 and 7. The total score is divided by 9 and if the mean is <4, it is assessed as no fatigue, if >4, it is assessed as fatigue. The FSS Turkish form, which has been validated and validated as reliable, will be used.
Assessment of Quality of Life | At baseline and after 12 weeks of exercise training
  Quality of life will be assessed using the 30-item European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ30). The EORTC QLQ-C30 is a valid and reliable cancer-specific quality of life scale. The scale includes three subheadings and 30 questions: general health, functional and symptom scales. In the first 28 questions showing the functional and symptom scales, there are four-point Likert options for each question: not at all (1 point), a little (2 points), quite a bit (3 points), and a lot (4 points). In the 29th question of the scale, the patient is asked to score their health from 1 to 7 (1: very poor and 7: excellent); and in the 30th question, they are asked to evaluate their general quality of life. The scores obtained from all questions of the scale range from 0 to 100 points.

CONTACTS AND LOCATIONS:
Overall Officials: Didem Karadibak, PhD, Principal Investigator — Dokuz Eylul University, Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No